CLINICAL TRIAL: NCT02767089
Title: A Randomized, Single-blind, Placebo-controlled, Crossover Studyto Assess The Dose Response Of Prednisone On Biochemical Andclinical Markers Of Efficacy And Safety In Adult Healthyvolunteers
Brief Title: The Dose Response of Prednisone on Biochemical and Clinical Makers in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: A9001309
Record Dates: First submitted 2016-04-21; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Adults
Keywords: Glucocorticoids, Biomarkers, Dissociated Agonist of the Glucocorticoid Receptor
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Sequence A (Other): Period 1: Placebo Period 2: Prednisone 2.5 mg Period 3: Prednisone 10 mg
  Interventions: Drug: Prednisone; Drug: Placebo
- Sequence B (Other): Period 1: Prednisone 2.5 mg Period 2: Prednisone 5 mg Period 3: Prednisone 20 mg
  Interventions: Drug: Prednisone
- Sequence C (Other): Period 1: Prednisone 5 mg Period 2: Prednisone 10 mg Period 3: Prednisone 40 mg
  Interventions: Drug: Prednisone
- Sequence D (Other): Period 1: Prednisone 10 mg Period 2: Prednisone 20 mg Period 3: Prednisone 60 mg
  Interventions: Drug: Prednisone
- Sequence E (Other): Period 1: Prednisone 20 mg Period 2: Prednisone 40 mg Period 3: Placebo
  Interventions: Drug: Prednisone; Drug: Placebo
- Sequence F (Other): Period 1: Prednisone 40 mg Period 2: Prednisone 60 mg Period 3: Prednisone 2.5 mg
  Interventions: Drug: Prednisone
- Sequence G (Other): Period 1: Prednisone 60 mg Period 2: Placebo Period 3: Prednisone 5 mg
  Interventions: Drug: Prednisone; Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — Subjects will receive oral prednisone and/or placebo tablets (total of 4 tablets) to achieve the required dose according to the treatment sequence group they were randomized. Subjects are to be dosed each morning for 7 days. A 14 day washout period is required between each period. Prednisone was supplied in the 2.5 and 20 mg dosage strengths.
Drug: Placebo — Placebo tablets similar to Prednisone 2.5 mg and 20 mg were supplied to make the trial doses.
  Arms: Sequence A; Sequence E; Sequence G

SUMMARY:
The purpose of this study is to further access the utility of biochemical and clinical biomarkers for glucocorticoid-mediated anti-inflammatory effects and safety endpoints against which dissociated agonists of the glucocorticoid receptor (DAGR) will be evaluated in adult healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females willing to be confined and comply with scheduled visits
* Women are to be surgically sterile.

Exclusion Criteria:

* History of febrile illness within 5 days prior to the first dose
* Positive urine drug screen
* Treatment with an investigational product within 30 days prior to the first dose of study medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on osteocalcin | 8 days
  The change in serum osteocalcin from baseline after treatment on Day 1 and Day 8 will be assessed in each treatment period
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on Cortisol Suppression | 8 days
  Change from baseline in serum cortisol after treatment on Day 1 and Day 8 in each treatment period
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on HPA Axis Suppression | 14 days after the last study visit in Period 3, if repeat testing required will be done 28 days after first test
  Serum cortisol in response to low-dose ACTH Stimulation Test will be completed at the end of Period 3 for each subject
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on White Blood Cell Counts | 8 days
  Change from baseline in blood leukocytes (neutrophils, lymphocytes and eosinophils) in each treatment period
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on Procollagen type 1-N-Propeptide (P1NP) | 8 days
  The change from baseline in serum P1NP after treatment on Day 1 and Day 8 will be assessed in each treatment period
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on Urinary N-terminal cross-linked telopeptide of type 1 collagen (uNTX-1) | 8 days
  Change from baseline in uNTX-1 will be assessed on Day 1 and Day 8 after treatment in each treatment period
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on Fasting glucose and insulin | 8 days
  Glucose and insulin will be assessed for the change from baseline after 7 days of treatment on Day 8 in each treatment period
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on an Oral Glucose Tolerance Test | Day 6
  On Day 6 of each period, subjects will undergo an oral glucose tolerance test. After ingesting 75 g of a glucose solution within 5 minutes of receiving their daily dose of prednisone, blood samples for glucose were obtained at 0.5, 1 and 2 hours.
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on Triglycerides | 8 days
  Change from baseline in triglycerides will be assessed after 7 days of treatment on Day 8 in each treatment period
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on Urinary Cortisol Suppression | 7 days
  Change from baseline in 24-hour urinary cortisol on Day 7 in each treatment period
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on Adiponectin | 8 days
  Change from baseline in adiponectin will be assessed after 7 days of treatment on Day 8 in each treatment period

SECONDARY OUTCOMES:
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on Profile of Mood State | 7 days
  Change from baseline after 7 days of treatment in each treatment period. The POMS is a copyrighted questionnaire that measures 6 dimensions of mood. The subject will assess how 65 descriptors apply to him/her on a 5-point scale of 0 (not at all) to 4 (extremely).
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on Medical Outcomes: Sleep Scale (MOS-Sleep) | 7 days
  Change from baseline in sleep after 7 days of treatment will be assessed in each treatment period. The patient-reported questionnaire consists of 12 items that assesses the key constructs of sleep. Scores can range from 12-71 with higher number indicating more problems with sleep.
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on the Incidence of Adverse Events | 28 days after last dose of study medication in Period 3
  Subjects were monitored throughout the study and queried for adverse events
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on Blood Pressure | 8 days
  Blood pressure will be assessed for change from baseline after 7 days of treatment on Day 8 in each treatment period
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on Weight | 8 days
  A post-void weight will be collected on the morning of Day 1 and Day 8 to assess change from baseline during each treatment period.
Characterize the dose-response effect of prednisone 2.5, 5, 10, 20, 40 and 60 mg on pulse rate | 8 days
  Pulse rate will be assessed for change from baseline after 7 days of treatment on Day 8 in each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Jasper Clinic, Inc., Kalamazoo, Michigan, United States

REFERENCES:
- [Derived] Fleishaker DL, Mukherjee A, Whaley FS, Daniel S, Zeiher BG. Safety and pharmacodynamic dose response of short-term prednisone in healthy adult subjects: a dose ranging, randomized, placebo-controlled, crossover study. BMC Musculoskelet Disord. 2016 Jul 16;17:293. doi: 10.1186/s12891-016-1135-3. PMID 27424036